CLINICAL TRIAL: NCT04255758
Title: Academic Investigational Study of Acute Effects of Vigorous-intensity Aerobic Exercise on Glymphatic Flow in Healthy Adults
Brief Title: Acute Effects of Vigorous-intensity Aerobic Exercise on Glymphatic Flow in Healthy Adults
Acronym: GLYMREG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Ilkka Heinonen, Adjunct Professor, Department of Clinical Medicine, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: T6/2020
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Glymphatic System; Neurodegeneration
Keywords: glymphatic system; cerebral perfusion; aerobic exercise
MeSH Terms: conditions — Nerve Degeneration

STUDY DESIGN:
Intervention Model Description: Prospective interventional study model, all subjects undergo the same exercise intervention and results are compared to baseline values
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vigorous-intensity Aerobic Exercise (Experimental): Vigorous-intensity aerobic exercise, single intervention
  Interventions: Other: Cycle Ergometer Exercise

INTERVENTIONS:
Other: Cycle Ergometer Exercise — 25 minutes, 70% VO2max steady state cycle ergometry exercise

SUMMARY:
This study investigates changes in glymphatic flow in the brain acutely after vigorous-intensity steady-state aerobic exercise. Twenty subjects (10 male and 10 female) perform 25 minute submaximal cycle ergometry exercise and the changes in the glymphatic flow and cerebral perfusion are evaluated using a variety of MRI sequences (e.g. MREG).

DETAILED DESCRIPTION:
The glymphatic system is a drainage system for the brain to help maintain fluid balance and extract waste metabolites. Glymphatic system function (healthy glymphatic flow) may prevent accumulation of harmful substances and therefore slow down the onset of neurodegenerative diseases.

The hypothesis is, that glymphatic flow could be increased through exercise and enhanced cerebral arterial pulsality, which might explain some of the brain health benefits of exercise proven in epidemiological studies. This study indirectly investigates the acute changes in the glymphatic flow acutely after aerobic exercise using MREG that measures pulse wave propagation as an indirect surrogate marker for glymphatic flow.

Twenty healthy subjects (n=20, 10 male, 10 female, age 18-45 years) will perform 25 minute 70%VO2max cycle ergometry exercise. The glymphatic flow and cerebral perfusion will be measured using magnetic resonance imaging sequences before and after exercise. The glymphatic flow is measured using 10 Hz fMRI technique called magnetic resonance encephalography (MREG). In addition, perfusion MRI is used to evaluate changes in brain perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* BMI 18-30
* Resting Blood pressure < 140/90 mmHg

Exclusion Criteria:

* History of a cardiac event
* Insulin or medically treated diabetes
* Any chronic disease or condition that could create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results
* Presence of ferromagnetic objects that would make MR imaging contraindicated
* Claustrophobia
* Abundant use of alcohol
* Use of narcotics
* Smoking of tobacco or consuming snuff tobacco
* Diagnosed depressive or bipolar disorder
* Abnormalities in resting ECG (revised by the study physician)
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
MREG cardiovascular pulse wavefront | 3 hours
  Is processed into three-dimensional vector fields and used as an assessment of glymphatic flow, scanned once before and multiple times after exercise intervention in 5-minute sequences

SECONDARY OUTCOMES:
Cerebral perfusion fMRI | 3 hours
  5-minute MR imaging sequences evaluating changes in blood flow, scanned once before and multiple times after exercise intervention
Heart rate (HR) | 3 hours
  Wearable heart rate monitoring, measures heart beats per second, continuous throughout the study
Blood pressure (BP) | 3 hours
  Blood pressure monitoring, evaluates systolic and diastolic pressures (mmHg) continuous throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka Heinonen, PhD, Principal Investigator — Turku PET Centre
Locations (1):
- Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajna Z, Raitamaa L, Tuovinen T, Heikkila J, Kiviniemi V, Seppanen T. 3D Multi-Resolution Optical Flow Analysis of Cardiovascular Pulse Propagation in Human Brain. IEEE Trans Med Imaging. 2019 Sep;38(9):2028-2036. doi: 10.1109/TMI.2019.2904762. Epub 2019 Mar 15. PMID 30892202
- [Background] von Holstein-Rathlou S, Petersen NC, Nedergaard M. Voluntary running enhances glymphatic influx in awake behaving, young mice. Neurosci Lett. 2018 Jan 1;662:253-258. doi: 10.1016/j.neulet.2017.10.035. Epub 2017 Oct 25. PMID 29079431